CLINICAL TRIAL: NCT02339337
Title: A Randomized-Controlled, Comparative Study, To Evaluate the Efficacy of Tailored Regimen of Peginterferon Alfa Plus Ribavirin According to Rapid Virological Response and Baseline Viral Loads in the Treatment of Patients With Chronic Hepatitis C/Hepatitis B Co-Infection: A Pilot Study (Pioneer)
Brief Title: A Pilot Study To Evaluate the Efficacy of Response Guided Therapy of Peginterferon Alfa Plus Ribavirin in the Treatment of Patients With HCV/HBV Co-Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-980019
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: HBV/HCV Co-infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RGT group (Experimental): For subjects who were randomized into the RGT group, the duration of Peg-IFN and RBV therapy was abbreviated to 24 weeks in subjects with HCV genotype 1, a pre-treatment low viral load (LVL, < 400000 IU/mL) and RVR (defined asHCV RNA <50 IU/mL at 4th week of therapy); the duration was 16 weeks in subjects with HCV genotype 2/3 and RVR.
  Interventions: Other: Abbreviation of treatment duration
- GGT group (Active Comparator): Subjects who were randomized into the GGT group received Peg-IFN and standard dose RBV (1200 mg/day) for 48 weeks in subjects infected with HCV genotype 1 or Peg-IFN and low dose RBV (800 mg/day) for 24 weeks in subjects infected with HCV genotype 2/3; the patients were then followed for 6 months.
  Interventions: Other: Abbreviation of treatment duration

INTERVENTIONS:
Other: Abbreviation of treatment duration

SUMMARY:
This is an open label, randomized-controlled, comparative trial. HBV and HCV dually infected patients with negative hepatitis B e antigen (HBeAg) were enrolled in the study. The definition of HBV and HCV dual infection included seropositivity of HCV antibody (anti-HCV) and HBsAg for more than 6 months, together with positive serum HCV RNA. Eligible subjects were randomized into 2 groups at treatment initiation. Subjects who were randomized into the genotype guided therapy (GGT) group received Peg-IFN and standard dose RBV (1200 mg/day) for 48 weeks in subjects infected with HCV genotype 1 or Peg-IFN and low dose RBV (800 mg/day) for 24 weeks in subjects infected with HCV genotype 2/3; the patients were then followed for 6 months. For subjects who were randomized into the response guided therapy (RGT) group, the duration of Peg-IFN and RBV therapy was abbreviated to 24 weeks in subjects with HCV genotype 1, a pre-treatment low viral load (LVL, < 400000 IU/mL) and RVR (defined asHCV RNA <50 IU/mL at 4th week of therapy); the duration was 16 weeks in subjects with HCV genotype 2/3 and RVR.

ELIGIBILITY:
Inclusion Criteria:

* seropositivity of HCV antibody (anti-HCV) and HBsAg for more than 6 months, together with positive serum HCV RNA.
* negative HBeAg
* serum alanine aminotransferase (ALT) levels between 1-10-fold of the upper limit of normal (ULN)
* treatment naive or had previously failed interferon monotherapy.

Exclusion Criteria:

* decompensated liver disease (Child-Pugh score ≥ 7)
* Pregnant or breast-feeding women
* serum creatinine ≥ 2 mg/dL
* evidence of alcoholism or drug abuse
* any other known disease that was not suitable for Peg-IFN therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of HCV sustained virological response | 6 months after completion of therapy